CLINICAL TRIAL: NCT01524159
Title: Bromelain and Cardiovascular Risk Factors in Diabetes
Acronym: BRCARDIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebei Yiling Hospital (Other)
Collaborators: London South Bank University (Other)
Responsible Party: Principal Investigator, Ley Chit Moy (Kara), PhD student, Hebei Yiling Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BR2012
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-01

CONDITIONS: Cardiovascular Disease.
Keywords: cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Bromelains

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo group (Placebo Comparator): This group will receive placebo capsule (wheat starch) for 12 weeks period. The 1050 mg dosage of wheat starch was divided into three capsules and to be taken two (2 x 350 mg) after breakfast and another one (350 mg) after dinner. The capsules should be taken two hours after the meals.
  Interventions: Dietary Supplement: placebo (wheat starch)
- bromelain group (Active Comparator): Bromelain Group This group will receive bromelain capsule for 12 weeks period. The 1050 mg dosage of bromelain was divided into three capsules and to be taken two (2 x 350 mg) after breakfast and another one (350 mg) after dinner. The capsules should be taken two hours after the meals.
  Interventions: Dietary Supplement: bromelain capsule

INTERVENTIONS:
Dietary Supplement: bromelain capsule — Bromelain group received bromelain capsule for 12 weeks period. The 1050 mg dosage of bromelain was divided into three capsules and to be taken two (2 x 350 mg) after breakfast and another one (350 mg) after dinner. The capsules should be taken two hours after the meals.
  Arms: bromelain group
Dietary Supplement: placebo (wheat starch) — Placebo group received placebo capsule (wheat starch) for 12 weeks period. The 1050 mg dosage of wheat starch was divided into three capsules and to be taken two (2 x 350 mg) after breakfast and another one (350 mg) after dinner. The capsules should be taken two hours after the meals.
  Arms: placebo group

SUMMARY:
The purpose of the study is to evaluate the effect of dietary supplementation of bromelain (a proteolytic enzyme from the pineapple plant) on the reduction of plasma fibrinogen level among type 2 diabetic subjects who have a high risk of cardiovascular disease.

The null hypothesis [Ho] is: there is no significant improvement in plasma fibrinogen, serum lipid profile, blood pressure, BMI, waist circumference and C-reactive protein for subjects with type 2 diabetes who are at risk of CVD following the intervention of bromelain supplementation compared to placebo group.

The alternative hypothesis [H1] is: there is a significant improvement in plasma fibrinogen, serum lipid profile, blood pressure, BMI, waist circumference and C-reactive protein for subjects with type 2 diabetes who are at risk of CVD following the intervention of bromelain supplementation compared to placebo group.

DETAILED DESCRIPTION:
According to American Heart Association (2010), heart disease and stroke are the No. 1 causes of death and disability among people with type 2 diabetes. At least 65% of people with diabetes die from some form of heart disease or stroke. Type 2 diabetes is associated with a two to fourfold increased incidence of ischemic cardiovascular events and markedly enhances the risk of stroke(Coutinho et al, 1999) due to a variety of associated risk factors that include high blood pressure, lipid disorders, high low-density lipoproteins (LDL) cholesterol, high triglycerides, low high-density lipoproteins (HDL) cholesterol, smoking, obesity, lack of physical activity and poorly controlled blood sugars(American Heart Association 2010).

Bromelain, a crude extract from the pineapple plant, was first introduced as a therapeutic compound in 1957 (Heinicke & Gortner, 1957). Heinicke et al. (1971) reported that bromelain was effective for use in cardiovascular diseases as an inhibitor of blood platelet aggregation, minimizing the risk of arterial thrombosis and embolism.

A literature review identified only three human studies (in Honolulu and Germany). In view of this review and the valuable therapeutic properties of bromelain to cardiovascular disease, there is a need for a study to confirm bromelain's use for cardiovasular disease.

This study is a randomized placebo control, parallel design, and double blind, pilot efficacy study which was carried out in Hebei Yiling Hospital, China. The study assessed the effects of 12 weeks of bromelain (1050mg/day) supplementation on plasma fibrinogen level compared to usual care. Study participants were type 2 diabetes who have a risk of developing cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years old
* Diagnosed type 2 diabetes (HbA1C at >6,5%), who are at a risk of CVD indicated with the following risk parameters:

  * total cholesterol between 5.0 - 6.2 mmol/l (195.0 - 241.8 mg/dL),
  * Body Mass Index (BMI) > 25 kg/m2
  * Waist circumference > 101.6 cm (40 inches) for men and > 88.9 cm (35 inches) for women
  * Triglycerides > 1.7 mmol/L (150mg/dL)
  * HDL-cholesterol < 1 mmol/L (40 mg/dL) for men, < 1.3 mmol/L (50 mg/dL) for women
  * LDL-cholesterol > 2.6 mmol/L (100 mg/dL)
  * Blood pressure > 140/90mm Hg

Exclusion Criteria:

* Pregnant or trying to become pregnant or lactating women
* Subjects unwilling or unable to comply with study procedure
* Subjects with severe health problems including renal disease, liver disease, cardiovascular disease, and other chronic ill health conditions.
* Subjects on drug cardiovascular medication like warfarin, aspirin.
* Subjects that are taking statins.
* Subjects taking bromelain supplement and other herbal supplements known to be effective e.g. cinnamon.
* Subjects have a history of allergic reactions to bee stings, olive tree pollen or pineapple.
* Subjects have a history of occupational inhalant/skin contact with bromelain.
* Subjects have diabetes ketoacidosis recently (past 2 weeks).
* Unable to provide informed consent i.e. unable to follow diet control advice or not willing to follow study procedure.
* Subjects who is on any Chinese herbs medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
fibrinogen | 12 weeks
  This study is to assess the effects of 12 weeks of bromelain (1050mg/day) supplementation on plasma fibrinogen level compared to usual care.

SECONDARY OUTCOMES:
Serum lipid profile (total cholesterol, HDL-cholesterol, LDL-cholesterol and triglycerides) | 12 weeks
  This study is to assess the effects of 12 weeks of bromelain (1050mg/day) supplementation on changes of serum lipid profile compared to usual care.
HbA1c | 12 weeks
  This study is to assess the effects of 12 weeks of bromelain (1050mg/day) supplementation on changes of HbA1c compared to usual care.
C-reactive protein | 12 weeks
  This study is to assess the effects of 12 weeks of bromelain (1050mg/day) supplementation on changes of C-reactive protein compared to usual care.
Body Mass Index | 12 weeks
  This study is to assess the effects of 12 weeks of bromelain (1050mg/day) supplementation on changes of body mass index compared to usual care.
Blood pressure | 12 weeks
  This study is to assess the effects of 12 weeks of bromelain (1050mg/day) supplementation on changes of blood pressure compared to usual care.
Alanine transaminase | 12 weeks
  This study is to assess the effect of 12 weeks of bromelain (1050mg/day) supplementation on changes of alanine transaminase (for liver function test) compared to usual care.
Aspartate aminotransferase | 12 weeks
  This study is to assess the effect of 12 weeks of bromelain (1050mg/day) supplementation on changes of aspartate aminotransferase(for liver function test) compared to usual care.
blood urea nitrogen | 12 weeks
  This study is to assess the changes of 12 weeks of bromelain (1050mg/day) supplementation on blood urea nitrogen(for kidney function test) compared to usual care.
Creatinine | 12 weeks
  This study is to assess the effect of 12 weeks of bromelain (1050mg/day) supplementation on changes of creatinine(for kidney function test) compared to usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Ley C M, Ms, Principal Investigator — London South Bank University
Locations (1):
- Hebei Yiling Hospital, Shijiazhuang, Beijing Municipality, China

REFERENCES:
- [Background] American Heart Association. Prevention, Secondary. 2010. Available online at www.americanheart.org/print_presenter.jhtml [assessed 17th April 2010]
- [Background] Heinicke, R.M. & Gortner, W.A. 1957. Stem Bromelain - A New Protease Preparation from Pineapple Plants. Economic Botany, 11, 225-234
- [Background] Heinicke RM, van der Wal L, Yokoyama M. Effect of bromelain (Ananase) on human platelet aggregation. Experientia. 1972 Jul 15;28(7):844-5. doi: 10.1007/BF01923166. No abstract available. PMID 4658882
- [Background] Coutinho M, Gerstein HC, Wang Y, Yusuf S. The relationship between glucose and incident cardiovascular events. A metaregression analysis of published data from 20 studies of 95,783 individuals followed for 12.4 years. Diabetes Care. 1999 Feb;22(2):233-40. doi: 10.2337/diacare.22.2.233. PMID 10333939